CLINICAL TRIAL: NCT01066923
Title: Enhanced Firefighter Rehab Trial: Aspirin Versus Placebo
Brief Title: Enhanced Firefighter Rehab Trial: The Role of Aspirin in Preventing Heat Stress Induced Platelet Activation
Acronym: EFFoRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dave Hostler (Other)
Collaborators: Federal Emergency Management Administration (Unknown); Eyemarker Systems, Inc (Industry)
Responsible Party: Sponsor-Investigator, Dave Hostler, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMW-2008-FP-01638
Record Dates: First submitted 2010-02-05; First posted 2010-02-10 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Heat Stress Disorders
Keywords: firefighter; heat stress; platelet activation; aspirin
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Daily ASA, Active cool, Acute ASA (Experimental): Two weeks of daily aspirin therapy prior to exercise, active cooling following exercise, aspirin immediately post exercise
  Interventions: Drug: Daily aspirin (ASA); Other: Active cooling; Drug: Acute aspirin (ASA)
- Daily ASA, Active cool, Acute placebo (Experimental): Two weeks of daily aspirin therapy prior to exercise, active cooling following exercise, placebo immediately post exercise
  Interventions: Drug: Daily aspirin (ASA); Other: Active cooling; Drug: Acute placebo
- Daily ASA, Passive cool, Acute ASA (Experimental): Two weeks of daily aspirin therapy prior to exercise, passive cooling following exercise, aspirin immediately post exercise
  Interventions: Drug: Daily aspirin (ASA); Drug: Acute aspirin (ASA); Other: Passive cooling
- Daily ASA, Passive cool, Acute placebo (Experimental): Two weeks of daily aspirin therapy prior to exercise, passive cooling following exercise, placebo immediately post exercise
  Interventions: Drug: Daily aspirin (ASA); Other: Passive cooling; Drug: Acute placebo
- Daily placebo, active cool, Acute ASA (Experimental): Two weeks of daily placebo prior to exercise, active cooling following exercise, aspirin immediately post exercise
  Interventions: Other: Active cooling; Drug: Acute aspirin (ASA); Drug: Daily placebo
- Daily placebo, active cool, Acute placebo (Experimental): Two weeks of daily placebo prior to exercise, active cooling following exercise, placebo immediately post exercise
  Interventions: Other: Active cooling; Drug: Daily placebo; Drug: Acute placebo
- Daily placebo, Passive cool, Acute ASA (Experimental): Two weeks of daily placebo prior to exercise, passive cooling following exercise, aspirin immediately post exercise
  Interventions: Drug: Acute aspirin (ASA); Other: Passive cooling; Drug: Daily placebo
- Daily placebo, Passive cool, Acute placebo (Placebo Comparator): Two weeks of daily placebo prior to exercise, passive cooling following exercise, placebo immediately post exercise
  Interventions: Other: Passive cooling; Drug: Daily placebo; Drug: Acute placebo

INTERVENTIONS:
Drug: Daily aspirin (ASA) — Two weeks 82 mg aspirin taken orally prior to exercise protocol
  Arms: Daily ASA, Active cool, Acute ASA; Daily ASA, Active cool, Acute placebo; Daily ASA, Passive cool, Acute ASA; Daily ASA, Passive cool, Acute placebo
Other: Active cooling — Active cooling to remediate heat stress following exercise by placing hands and forearms into cold water
  Arms: Daily ASA, Active cool, Acute ASA; Daily ASA, Active cool, Acute placebo; Daily placebo, active cool, Acute ASA; Daily placebo, active cool, Acute placebo
Drug: Acute aspirin (ASA) — 325 mg chewable aspirin administered immediately following exercise
  Arms: Daily ASA, Active cool, Acute ASA; Daily ASA, Passive cool, Acute ASA; Daily placebo, Passive cool, Acute ASA; Daily placebo, active cool, Acute ASA
Other: Passive cooling — Removing protective garments for passive cooling following exercise
  Arms: Daily ASA, Passive cool, Acute ASA; Daily ASA, Passive cool, Acute placebo; Daily placebo, Passive cool, Acute ASA; Daily placebo, Passive cool, Acute placebo
Drug: Daily placebo — Placebo comparator for daily aspirin therapy
  Arms: Daily placebo, Passive cool, Acute ASA; Daily placebo, Passive cool, Acute placebo; Daily placebo, active cool, Acute ASA; Daily placebo, active cool, Acute placebo
Drug: Acute placebo — Placebo comparator for acute aspirin therapy
  Arms: Daily ASA, Active cool, Acute placebo; Daily ASA, Passive cool, Acute placebo; Daily placebo, Passive cool, Acute placebo; Daily placebo, active cool, Acute placebo

SUMMARY:
The purpose of this study is to determine if aspirin taken by firefighters prevents platelets from becoming sticky when body temperature rises during work in protective clothing.

DETAILED DESCRIPTION:
Firefighters have the highest rate of line-of duty death (LODD) in the United States. More than half of these LODD are cardiovascular related occurring disproportionately around fire suppression activities. In addition, shift work, lifestyle factors, and the exposures associated with fire suppression (e.g. smoke, chemicals) may predispose the firefighter to earlier onset of heart disease or cause a pro-inflammatory state leading to endothelial dysfunction.

Fire suppression activities exacerbate cardiovascular strain and endothelial dysfunction and provide potential triggers for ischemic events (e.g. myocardial infarction, stroke). There is a rapid rise in heart rate following the activation of a fire company which may persist for as long as 20 minutes. Even in cases where heavy work is not being performed, the repetitive upper body exercise associated with tool use raises heart rate disproportionately to oxygen consumption.

Finally, there is a rapid rise in core body temperature from increased physical activity, environmental heat and impaired thermoregulation that has been shown to cause vasoconstriction and activate coagulation during heat stress (12, 13). This has recently been demonstrated in firefighters working in thermal protective clothing. The combination of triggers created during fire suppression may result in heart attack or stroke, especially in firefighters with risk factors for cardiovascular disease.

Interventions beyond basic fireground rehab may be required to minimize the effect of these triggers and enhance a firefighter's health and wellness. Fireground rehab typically focuses on cooling and rehydration of the firefighter following fire suppression or training with the assumption that these interventions will correct the underlying pathophysiology. Effective fireground rehab must deliver appropriate interventions and monitor the progress of the firefighter. While correcting hyperthermia and hypohydration are essential for continued performance, it is not clear if these therapies correct alterations in platelet or endothelial function or if other interventions are necessary to correct these physiological disturbances. Furthermore, the options for monitoring the firefighter beyond simply measuring heart and respiratory rate are limited. In our FEMA-funded Fireground Rehab Evaluation (FIRE) Trial, we demonstrated that five commercially available thermometers did not reliably measure or estimate core temperature following uncompensable heat stress (UHS) making it impossible to gauge the effectiveness of rehab interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy males and females aged 18-49 years

Exclusion Criteria:

1. History of heart disease, vascular disease, or sudden death including prior MI, coronary revascularization, congenital heart disease or history of stroke
2. Hypertension during screening: SBP>139 or DBP>89
3. Those who are taking medications that may be expected to blunt the physiologic response to a treadmill exercise test (e.g. beta blockers)
4. Prescription medication with known side effect of impaired thermoregulation
5. Positive pregnancy test at any time during the study
6. Resting ECG with clinical presentation suggesting coronary heart disease (e.g. pathologic Q wave)
7. Known history of gastrointestinal disease or disorder i.e. diverticulitis which creates a theoretical risk of the core temperature capsule becoming lodged in the digestive tract
8. Medications and supplements known to alter endothelial function (e.g. arginine, omega 3 fatty acids, NSAIDS, tobacco products. This exclusion may be disregarded for subjects willing to stop taking the supplement for the duration of the study
9. At the discretion of the study physician for any other medical condition or prescription medication
10. Known history of platelet dysfunction
11. Aspirin allergy or intolerance

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hostler, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Emergency Responder Human Performance Lab, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Olafiranye O, Hostler D, Winger DG, Wang L, Reis SE. Effect of aspirin on acute changes in peripheral arterial stiffness and endothelial function following exertional heat stress in firefighters: The factorial group results of the Enhanced Firefighter Rehab Trial. Vasc Med. 2015 Jun;20(3):230-6. doi: 10.1177/1358863X15571447. Epub 2015 May 4. PMID 25939657
- [Result] Hostler D, Suyama J, Guyette FX, Moore CG, Pryor RR, Khorana P, McEntire SJ, Comer D, Reis SE. A randomized controlled trial of aspirin and exertional heat stress activation of platelets in firefighters during exertion in thermal protective clothing. Prehosp Emerg Care. 2014 Jul-Sep;18(3):359-67. doi: 10.3109/10903127.2013.869644. Epub 2014 Feb 18. PMID 24548114
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/25939657 — Report of vascular function testing
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/24548114 — Report of platelet function and physiology

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Active Cooling Arm not completed - insufficient number of subjects were recruited to complete these arms of the trial, and the Passive Cooling arms were the only ones conducted.
Period: Overall Study
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo
Started | 28 | 32 | 33 | 31
Platelet Closure Time | 25 | 29 | 25 | 23
Vascular Function | 13 | 14 | 12 | 13
Activation of Coagulation | 0 | 0 | 0 | 0
Retinal Imaging | 0 | 0 | 0 | 0
Completed | 25 | 29 | 25 | 23
Not Completed | 3 | 3 | 8 | 8
Not completed — Withdrawal by Subject | 3 | 3 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo | Total
Number analyzed (Participants) | 25 | 29 | 25 | 23 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.1) | 29.3 (8.6) | 30.5 (8.5) | 34.5 (9.3) | 31.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 0 | 8
  Male | 24 | 26 | 21 | 23 | 94
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 25 | 23 | 102

OUTCOME MEASURES:

1. Primary Outcome: Platelet Closure Time
Time Frame: 0, 30, 60, and 90 minutes post exercise
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo
Number analyzed (Participants) | 25 | 29 | 25 | 23
seconds
  Immediate post exercise | 275.5 [62 to 300] | 207 [55 to 300] | 95 [71 to 182] | 90 [58 to 201]
  30 minutes post | 300 [300 to 300] | 300 [150 to 300] | 300 [110 to 300] | 105 [80 to 120]
  60 minutes post | 300 [300 to 300] | 300 [120 to 300] | 300 [125 to 300] | 105 [80 to 120]
  90 minutes post | 300 [300 to 300] | 275 [120 to 300] | 300 [150 to 300] | 105 [80 to 120]

2. Primary Outcome: Vascular Function Measured by Peripheral Arterial Tonometry
Description: Reactive Hyperemia Index
Time Frame: Baseline, 30, 60, and 90 minutes post exercise
Measure: Mean (Standard Deviation); unit: ratio (Reactive Hyperemia Index)
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo
Number analyzed (Participants) | 13 | 14 | 12 | 13
ratio (Reactive Hyperemia Index)
  Baseline | 1.89 (0.38) | 1.77 (0.51) | 2.16 (0.74) | 1.72 (0.34)
  30 minutes post | 1.97 (0.56) | 1.77 (0.38) | 1.77 (0.71) | 1.73 (0.30)
  60 minutes post | 2.18 (0.48) | 1.92 (0.48) | 1.56 (0.68) | 1.83 (0.40)
  90 minutes post | 2.09 (0.31) | 1.98 (0.45) | 1.91 (0.66) | 1.98 (0.51)

3. Secondary Outcome: Activation of Coagulation
Description: This measure was not collected. Equipment was not available.
Time Frame: 0, 30, 60, and 90 minutes post exercise
Population: This measure was not collected. Equipment was not available.
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Hyperthermia and Hemoconcentration Identified by Retinal Imaging
Description: This measure was not collected. Equipment was not available.
Time Frame: 0, 30, 60, and 90 minutes post exercise
Population: This measure was not collected. Equipment was not available.
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Daily ASA, Passive Cool, Acute ASA | Daily ASA, Passive Cool, Acute Placebo | Daily Placebo, Passive Cool, Acute ASA | Daily Placebo, Passive Cool, Acute Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/29 | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/29 | 0/25 | 0/23

LIMITATIONS AND CAVEATS:
Detailed results at Olafiranye et al. (2015) Vascular Medicine 20:230-236 and at Hostler et al. (2014) Prehospital Emergency Care 18: 359-367 These papers are linked in the Reference Section

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No